CLINICAL TRIAL: NCT03102333
Title: Comparison: Constant-rate Infusion Plus Demanding Dosing VS Variable-rate
Brief Title: Comparison: Constant-rate Infusion Plus Demanding Dosing VS Variable-rate Feedback Infusion Plus Demanding Dosing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Chongwha Baek, Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CAUH-SP1
Record Dates: First submitted 2017-03-08; First posted 2017-04-05 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Constant-rate Infusion (Active Comparator): INTERVENTION : Constant-rate Infusion mode : The PCA regimen consisted of fentanyl 20 μg/kg and Ramosetron Hcl 0.3 mg (total volume including saline: 100 ml) and was programmed to deliver 1 ml /h as a background infusion and a bolus of 1.5 ml on-demand, with a 15 min lockout time during a 48 h period
  Interventions: Device: Constant-rate Infusion mode
- Variable-rate Feedback Infusion (Active Comparator): INTERVENTION : Variable-rate Feedback Infusion mode :The PCA regimen consisted of fentanyl 20 μg/kg and Ramosetron Hcl 0.3 mg (total volume including saline: 100 ml) and was programmed to deliver 1 ml /h as a background infusion and a bolus of 1.5 ml on-demand, with a 15 min lockout time. It can increment or decrement rate(0.2ml/hr) by press bolus button during a 48 h period
  Interventions: Device: Variable-rate Feedback Infusion mode

INTERVENTIONS:
Device: Variable-rate Feedback Infusion mode — The PCA regimen consisted of fentanyl 20 μg/kg and Ramosetron Hcl 0.3 mg (total volume including saline: 100 ml) and was programmed to deliver 1 ml /h as a background infusion and a bolus of 1.5 ml on-demand, with a 15 min lockout time. It can increment or decrement rate(0.2ml/hr) by press bolus button during a 48 h period
  Arms: Variable-rate Feedback Infusion
Device: Constant-rate Infusion mode — The PCA regimen consisted of fentanyl 20 μg/kg and Ramosetron Hcl 0.3 mg (total volume including saline: 100 ml) and was programmed to deliver 1 ml /h as a background infusion and a bolus of 1.5 ml on-demand, with a 15 min lockout time during a 48 h period
  Arms: Constant-rate Infusion

SUMMARY:
In the case of the newlys developed PCA, the infusion rate is increased according to the patient's need for bolus button, so that the pain can be controlled more efficiently.

DETAILED DESCRIPTION:
In the case of the existing iv-pca, the analgesic drug was injected into the patient at a constant rate (ex. 1 ml / hr) and additional pain was controlled through the bolus dose (1 ml).

As a result, the analgesic effect was insufficient, or the effect was excessive, causing side effects (nausea, vomiting, sedation, dizziness). Especially In spinal surgery, the degree of pain sharply decreases from day 1 to day 2. Classic iv-pca with constant infusion rate can not reflect this result. But in the case of the newlys developed PCA, the infusion rate is increased according to the patient's need for bolus button, so that the pain can be controlled more efficiently. If the bolus button is not pressed for a certain period of time, it is expected that the injection rate will be reduced and the side effect caused by the analgesic agent will be decreased.

ELIGIBILITY:
Inclusion Criteria:

* Spine fusion surgery at Chung-Ang University Hospital with IV- PCA under general anesthesia

Exclusion Criteria:

* Unrecorded type of anesthetic agent
* Denial to the study
* Brain disorder
* Cardiopulmonary disease
* Psychiatric disorders

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Demanded numbers of bolus button | Change from immediately to 24 hours after operation

SECONDARY OUTCOMES:
Pain intensity | Change from immediately to 24 hours after operation
  by Numerical Rating Scale(NRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided